CLINICAL TRIAL: NCT02544997
Title: A Phase II, Single-Arm Trial of Poziotinib as Salvage Treatment in Patients With Metastatic Breast Cancer Who Has HER2 or EGFR Mutation or Activated AR or EGFR Pathway
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-11-078
Record Dates: First submitted 2015-09-06; First posted 2015-09-09 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Poziotinib (Experimental): 12mg P.O. for 2wks q21days
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — 12mg P.O. for 2wks q21days
  Other Names: HM781-36B

SUMMARY:
Metastatic breast cancer (MBC) is an incurable disease and is needed to improve effective therapeutic strategies including targeted agents.

Poziotinib is a panHER tyrosin kinase inhibitor (TKI) that showed stable activity with feasible toxicity for MBC patients as a salvage treatment strategy after failure of anthracycline and taxane in phase I trial. Poziotinib has rational benefit compared with other salvage agents, especially for patients with HER2 overexpression breast cancers. Additionally, a recent report showed that possible rational background for patients with HER2 mutation-positive breast cancers.

Based on this rationale, the investigators are to conduct phase II single-arm study of poziotinib for patients with MBC who showed refractoriness to conventional treatments as salvage treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic breast cancer with measurable or evaluable disease
2. age ≥ 20 years
3. HER2 mutation or EGFR mutation/gene amplification confirmed by CancerSCAN or Activated AR pathway confirmed by RNA seq & nCounter assay, AR expression was confirmed by immunohistochemistry(IHC) or EGFR high expression (≥ IHC 2+ & lower ER / ≥ IHC score + and HER2 2+ or SISH negative)
4. ECOG performance status 0 - 2
5. Two or more regimens for locally recurrent or metastatic breast cancer, including an anthracycline and a taxane
6. Life expectancy ≥ 3 months
7. Progression within 6 months or less of latest chemotherapy
8. The patients must have recovered from the acute toxic effects of the treatment prior to study enrollment. Prior radiotherapy must be completed 2 weeks before study entry.
9. Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
10. Adequate renal function (serum creatinine ≤ 1.5 x upper normal limit or CCr ≥ 50 ml/min)
11. Adequate liver function (serum bilirubin ≤ 1.5 x upper normal limit, AST/ALT ≤ 3 x upper normal limit)
12. No prior history of pan-HER TKI including poziotinib for metastatic breast cancer
13. Written informed consent

Exclusion Criteria:

1. HER2-overexpressing breast cancer
2. Serious uncontrolled intercurrent infections
3. Serious intercurrent medical or psychiatric illness, including active cardiac disease
4. Pregnancy or breast feeding
5. Second primary malignancy(except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin or resected thyroid papillary carcinoma or other malignancy treated at least 5 years previously with no evidence of recurrence)
6. Documented leptomeningeal brain metastasis
7. Known brain metastases unless treated and stable
8. Peripheral neuropathy ≥ grade 3
9. Prior treatment with pan-HER TKI including poziotinib will not be allowed.
10. Use of any investigational drug within 4 weeks of the study
11. Treatment with chemotherapy or hormone therapy within 3 weeks of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 years

SECONDARY OUTCOMES:
overall survival (OS) | 1 years
duration of response | 1 years
objective response rate | 1 years
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea